CLINICAL TRIAL: NCT00622180
Title: The Efficacy of Hand-Foot Narrow-Band Ultraviolet B (UVB) Versus Focal 308-nm Treatment in Inducing Repigmentation of Vitiligo After Minigrafting on the Dorsal Hands
Brief Title: The Efficacy of Hand Narrow-Band Ultraviolet B (NBUVB) Versus Excilite Treatment in Vitiligo After Minigrafting on the Dorsal Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB file number 122007-003; 122007-003
Record Dates: First submitted 2008-01-23; First posted 2008-02-22 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Vitiligo
Keywords: Vitiligo; Light treatment for vitiligo; Excilite
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daavlin Right vs. Excilite Left (Active Comparator): Right hand treated with narrow-band UVB light and left hand treated with focal 308nm light.
  Interventions: Device: NBUVB
- Excilite Right vs. Daavlin Left (Active Comparator): Right hand treated with focal 308-nm light and left hand treated with narrow-band UVB light
  Interventions: Device: Monochromacitc Excimer light

INTERVENTIONS:
Device: NBUVB — NBUVB hand foot box
  Arms: Daavlin Right vs. Excilite Left
Device: Monochromacitc Excimer light — Treatment with Monochromacitc Excimer light
  Arms: Excilite Right vs. Daavlin Left

SUMMARY:
To assess over a 25-week period the efficacy of hand-foot narrow-band ultraviolet B light versus focal 308-nm light treatment in inducing the return of pigment in vitiligo after skin minigraft transplants to the backs of the hands in patients with light brown to black skin. Subject will undergo treatment for 13 weeks.

DETAILED DESCRIPTION:
Prospective investigator-blinded study involving 13 adult male and female subjects with vitiligo on the backs of both hands. Punch minigrafting will be performed on both hands taking skin from the thighs and/or buttocks. Light treatments will be administered starting at week one after grafting. One hand will receive narrow-band ultraviolet B light and the other will receive focal 308-nm light treatments. Light treatments will be administered 3 times per week for 12 weeks. A long term follow-up visit will be completed at week 25. The investigator will evaluate the subjects at week 4, 7, 13 and 25 in addition to screening and baseline evaluations/procedures.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects 18 years of age or older
* skin type III-VI
* vitiligo on both dorsal hands
* history of stable vitiligo ( no new lesions and no more than 10% enlargement of existing lesions) for six months with an absence of Kebner phenomenon (new lesions appearing after trauma to the skin)
* refractory to topical steroids and immunomodulators

Exclusion Criteria:

* pregnant and/or breast-feeding females
* history of skin cancer
* history of taking photosensitizing medications
* history of recent phototherapy (light therapy) or topical medications within one month prior to enrollment
* history of organ transplantation
* history of failed vitiligo skin transplantation
* history of segmental vitiligo
* history of 12 or more continuous light treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Pandya, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas - Department of Dermatology
Locations (1):
- UT Southwestern Medical Center at Dallas - Dermatology Clinical Trials, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It was our hope to enroll 26 Participants but only 13 was enrolled.
Period: Overall Study
Arm/Group | Daavlin Right vs. Excilite Left | Excilite Right vs. Daavlin Left
Started | 6 | 7
Completed | 5 | 5
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- The Efficacy of Hand NBUVB Vs. Excilite Treatment in Vitiligo: Light therapy with the NBUVB hand-foot box to one hand and the Excilite to the other hand three times a week on non-consecutive days for a total of 12 weeks. The light will be dosed as follows: starting dose for NBUVB will be 200 mJ/cm2 with subsequent dose increases of 15% per treatment as tolerated. For the Excilite device, the starting dose will be 200 mJ with subsequent dose increases of 50 mJ per treatment as tolerated.
Arm/Group | The Efficacy of Hand NBUVB Vs. Excilite Treatment in Vitiligo
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Percent Repigmentation of Target Lesion
Description: This is measured using photography and Scion software calculations.
Time Frame: 25 weeks
Measure: Mean (Standard Deviation); unit: percentage of repigmentation
Groups:
- NBUVB: Treatment with NBUVB
- Monochromatic Excimer Light: One hand treated with monochromatic excimer light
Arm/Group | NBUVB | Monochromatic Excimer Light
Number analyzed (Participants) | 13 | 13
percentage of repigmentation | 0.21 (0.35) | 0.17 (0.38)

ADVERSE EVENTS:
Groups:
- Daavlin vs. Excilite: Right hand treated with narrow-band UVB light and left hand treated with focal 308nm light.
  Daavlin Spectra UVB Hand/Foot Box : Narrow-band ultraviolet B hand box
  Excilite Focal 308-nm light : Excilite Focal 308-nm light
- Excilite vs. Daavlin: Right hand treated with focal 308-nm light and left hand treated with narrow-band UVB light
  Excilite Focal 308-nm light : Excilite Focal 308-nm light
  Daavlin Spectra UVB Hand/Foot Box : Narrow-band ultraviolet B hand box
Arm/Group | Daavlin vs. Excilite | Excilite vs. Daavlin
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes